CLINICAL TRIAL: NCT04098874
Title: Bupropion for the Prevention of Postpartum Smoking Relapse
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMCH-2019-28219; R01DA047287 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Smoking Relapse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupropion (Experimental): Participants randomized to extended-release bupropion. Once-daily
  Interventions: Drug: Bupropion Extended Release Oral Tablet
- Placebo (Placebo Comparator): Participants randomized to placebo. Once-daily
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Bupropion Extended Release Oral Tablet — 12 weeks postpartum of blinded study medication
  Arms: Bupropion
Drug: Placebo oral tablet — 12 weeks postpartum of blinded placebo
  Arms: Placebo

SUMMARY:
This two-arm, double-blind, placebo-controlled randomized clinical trial will enroll pregnant women who quit smoking after learning they were pregnant and are motivated to stay abstinent postpartum. Participants will be randomized to receive extended-release bupropion (active 300mg or placebo once daily beginning 4 to 10 days postpartum to 12 weeks post-randomization). All participants will complete the same data collection procedures (e.g., biological sample collection for hormone and cotinine analysis and completion of validated questionnaires) at baseline (gestational week 36), weekly from 4 to 10 days postpartum through 12 weeks post-randomization and at weeks 12, 24, 36 and 52 post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Age 18 to 45 years old
* Stable health
* 7-day point prevalence abstinence demonstrated at randomization
* Lifetime history of at least 100 cigarettes smoked
* Quit smoking during the current pregnancy
* Self-report of intention to remain abstinent after delivery ≥ 7 on a 10 point Likert-type scale
* Uncomplicated delivery
* Denies plans to become pregnant again during the trial.
* Full-term delivery ≥ 37 weeks gestation
* Home within 10 days of delivery

Exclusion Criteria:

* Current use of other forms of tobacco or nicotine (e-cigs, chew, snuff, etc.)
* Current use of cessation aids (e.g., varenicline, NRT)
* Current use of illicit drugs or alcohol dependence
* Current use of antidepressant medication
* Bipolar disorder, eating disorder, or psychotic disorder based on the Structured Clinical Interview
* Medications & conditions that may increase the risk of taking bupropion (e.g., current or history of pulmonary embolus, stroke, heart disease, kidney disease, glaucoma, diabetes, seizure disorder, traumatic head injury, use of medications metabolized by CYP2D6)
* Family history of seizures or seizure disorder
* Maternal use of medications that lower seizure threshold
* Newborn with an elevated risk of seizure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals eligible for this study must be pregnant at the time of enrollment.
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Point prevalence smoking abstinence | 24 weeks post randomization
  7-day point prevalence abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Allen, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified data collected in this trial may be available to other researchers. Requests for data will be considered on an individual basis by the study team.

REFERENCES:
- [Derived] Allen S, Thomas J, Harrison K, Emery RL, Petersen A, Winickoff JP, Japuntich S. Bupropion for postpartum smoking relapse: A remote protocol for a two-arm, double-blind, placebo-controlled randomized clinical trial. Contemp Clin Trials. 2021 Jun;105:106352. doi: 10.1016/j.cct.2021.106352. Epub 2021 Mar 9. PMID 33706003